CLINICAL TRIAL: NCT01030211
Title: Adult Dengue Platelet Study
Acronym: ADEPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore General Hospital (Other); Changi General Hospital (Other); National University Hospital, Singapore (Other); University of Malaya (Other)
Responsible Party: Principal Investigator, David Lye, Dr David Lye, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTSH ADEPT
Record Dates: First submitted 2009-11-03; First posted 2009-12-11 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Dengue Fever
Keywords: Dengue; Platelet transfusion; Bleeding; Prevention
MeSH Terms: conditions — Dengue; Hemorrhage | interventions — Platelet Transfusion; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet transfusion (Active Comparator): 4 units of platelets for patients with platelet count <20x10^3/uL
  Interventions: Procedure: Platelet transfusion
- Supportive care (Other): No platelet transfusion for patients with platelet count <20x10^3/uL
  Interventions: Other: Supportive care

INTERVENTIONS:
Procedure: Platelet transfusion — 4 units of platelets for patients with platelet count <20x10^3/uL
  Arms: Platelet transfusion
Other: Supportive care — Supportive care includes symptomatic treatment, fluid therapy and monitoring of full blood count and blood pressure
  Arms: Supportive care

SUMMARY:
Retrospective data in children with dengue hemorrhagic fever (DHF) and dengue shock syndrome (DSS), and in adults with dengue fever (DF), suggested a lack of benefit from prophylactic platelet transfusion for severe thrombocytopenia in dengue patients without bleeding. However, in Taiwan and Singapore, platelet transfusion was given to 13-50% of hospitalised dengue patients. This is a prospective randomised study to examine the safety and efficacy of prophylactic platelet transfusion in adults with dengue and severe thrombocytopenia without bleeding.

The hypotheses are:

1. Prophylactic platelet transfusion is safe in hospitalised dengue patients with severe thrombocytopenia.
2. Prophylactic platelet transfusion is effective in preventing bleeding in hospitalised dengue patients with severe thrombocytopenia.

DETAILED DESCRIPTION:
Patients fulfilling inclusion and exclusion criteria, and giving informed consent, will be randomised to a treatment arm of 4 units of platelets for every day they have a platelet count <20x10^3/uL, or a control arm with supportive care. Patients will be followed up daily till hospital discharge, and again at day 21.

It is assumed that the incidence of bleeding from randomization to Day 7 or discharge, whichever earlier, is 10% for the control (no transfusion) group and 5% for the intervention (transfusion) group. With 1:1 allocation ratio, to attain 80% power and one-sided 5% type I error rate, the required number of subjects in each arm is 382 by a Chi-square test with Yates' continuity correction. If a drop-out rate of 5% is allowed, the required number increases to approximately 400 per arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21years
2. Probable or confirmed dengue

   a) Confirmed dengue: laboratory confirmation of acute dengue by either i) positive polymerase chain reaction (PCR) for viral ribonucleic acid (RNA), or ii)positive NS1 antigen test with a compatible clinical syndrome b) Probable dengue: Positive acute dengue serology and clinical presentation fulfilling either WHO 1997 or 2009 criteria for probable dengue.

   i) 1997 criteria: Acute febrile illness and two or more of the following:
   * headache,
   * retro-orbital pain,
   * myalgia,
   * arthralgia,
   * rash,
   * hemorrhagic manifestations,
   * leucopoenia ii) 2009 criteria: Fever and two of the following:
   * nausea/vomiting,
   * rash,
   * aches/pains,
   * positive tourniquet test,
   * leucopoenia,
   * one or more warning sign
   * abdominal pain/tenderness,
   * persistent vomiting,
   * clinical fluid accumulation,
   * mucosal bleed,
   * lethargy/restlessness,
   * liver enlargement >2cm,
   * increase in haematocrit concurrent with rapid decrease in platelet count
3. Platelets ≤ 20x103/μL

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Clinical bleeding excluding petechiae with a subgroup analysis for severe clinical bleeding. | 5 years

SECONDARY OUTCOMES:
Platelet increment post-transfusion | 5 years
Time to platelet > 50 x 10^3/uL | 5 years
Changes in cytokines | 5 years
Length of stay | 5 years
Plasma leakage | 5 years
DHF/DSS | 5 years
ICU admission | 5 years
Death | 5 years
Secondary bacterial infection | 5 years
Adverse events from transfusion | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yee S Leo, FRCP, Principal Investigator — Tan Tock Seng Hospital
Locations (2):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia
- Tan Tock Seng Hospital, National University Health System, Singapore General Hospital, Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Derived] Archuleta S, Chia PY, Wei Y, Syed-Omar SF, Low JG, Oh HM, Fisher D, Ponnampalavanar SSL, Wijaya L, Kamarulzaman A, Lum LCS, Tambyah PA, Leo YS, Lye DC. Predictors and Clinical Outcomes of Poor Platelet Recovery in Adult Dengue With Thrombocytopenia: A Multicenter, Prospective Study. Clin Infect Dis. 2020 Jul 11;71(2):383-389. doi: 10.1093/cid/ciz850. PMID 31626692
- [Derived] Lye DC, Archuleta S, Syed-Omar SF, Low JG, Oh HM, Wei Y, Fisher D, Ponnampalavanar SSL, Wijaya L, Lee LK, Ooi EE, Kamarulzaman A, Lum LC, Tambyah PA, Leo YS. Prophylactic platelet transfusion plus supportive care versus supportive care alone in adults with dengue and thrombocytopenia: a multicentre, open-label, randomised, superiority trial. Lancet. 2017 Apr 22;389(10079):1611-1618. doi: 10.1016/S0140-6736(17)30269-6. Epub 2017 Mar 8. PMID 28283286
- [Derived] Tomashek KM, Biggerstaff BJ, Ramos MM, Perez-Guerra CL, Garcia Rivera EJ, Sun W. Physician survey to determine how dengue is diagnosed, treated and reported in puerto rico. PLoS Negl Trop Dis. 2014 Oct 9;8(10):e3192. doi: 10.1371/journal.pntd.0003192. eCollection 2014 Oct. PMID 25299251